CLINICAL TRIAL: NCT02409784
Title: PET Study of Cerebral Metabolism of 11C-acetoacetate and 18F-FDG in Patients Under Moderate Ketosis
Acronym: TEP-KD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-214
Record Dates: First submitted 2015-03-27; First posted 2015-04-07 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Brain metabolism; Ketones; Ketogenic diet; TEP scan
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: Ten participants received a very high fat ketogenic diet (KD) (4.5:1; lipid:protein plus carbohydrates) for four days.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketogenic diet (Experimental): Pre/Post TEP study with a 4 days ketogenic diet (KD).
  Interventions 1: Pre-KD = Participants did a TEP before starting the 4-day diet
  Intervention 2: Post-KD = Participants did a TEP after completing the 4-day diet
  Interventions: Dietary Supplement: Pre-KD; Dietary Supplement: Post-KD

INTERVENTIONS:
Dietary Supplement: Pre-KD — Before starting 4 days of 4:1 (lipids:protein/carbohydrates) ketogenic diet
Dietary Supplement: Post-KD — After 4 days of 4:1 (lipids:protein/carbohydrates) ketogenic diet

SUMMARY:
Regional brain glucose hypometabolism occurs during aging and may contribute to the onset of aging-related cognitive impairment in humans. Ketones are the main alternative energy substrate to glucose for the brain. Several studies show that brain ketone uptake and metabolism are unaltered in cognitively-normal older persons and in Alzheimer's disease (AD). Nutritional ketosis is reported to have a positive impact on cognitive performances in mild cognitive impairment and AD. Nevertheless, changes in regional brain glucose and ketone uptake in adults are poorly understood during diet-induced experimental ketosis. The investigators hypothesis was that during diet-induced ketosis, brain ketone uptake would be directly correlated with the elevation of blood ketone levels and inversely correlated to brain glucose uptake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* No signs of cognitive impairment

Exclusion Criteria:

* Not within the age limits
* Pregnancy or breast feeding
* Incapacity to withstand a supine position for 40 min
* Non lacunar infarction
* Known psychiatric history of schizophrenia, psychotic disorders, major affective disorders (bipolar disorder and major depression <5 years), panic disorder, obsessive compulsive disorders and other conditions that may affect memory
* Epilepsy, brain trauma with loss of consciousness, subarachnoid hemorrhage
* History of alcool and/or substances abuse (excessive alcool consumption ≥10 drinks/weeks)
* Parkinson disease
* Down syndrome
* Inflammatory disease
* Abnormal blood pressure, liver or kidney function, blood count
* Dyslipidemia, hypothyroidism, osteoporosis
* Presence of a metal object in the body

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen C Cunnane, PhD, Principal Investigator — Université de Sherbrooke

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant were recruited with advertising poster on bulletin board of different local organism (university, health clinic, sport and leisure association, etc)
Groups:
- Ketogenic Diet: TEP study following a 4 day ketogenic diet (KD), consisting of a classic 4:1 KD (4:1 lipid to carbohydrate + protein ratio) in the form of liquid meal (water, cream, MCT oil, liquid egg white, flavor) and taken in 3 separates meal.
  Intervention 1: Pre-KD = Participants did a TEP before starting the 4 days ketogenic diet
  Intervention 2 : Post-KD = Participants did a TEP after the 4 days ketogenic diet
Period: Overall Study
Arm/Group | Ketogenic Diet
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ketogenic Diet: TEP study following a 4 day ketogenic diet (KD)
  Intervention 1: Pre-KD = Participants did a TEP before starting a 4 days ketogenic diet Intervention 2: Post-KD = Participants did a TEP after 4 days of ketogenic diet
Arm/Group | Ketogenic Diet
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  Canada | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean in Cerebral Metabolic Rate of Acetoacetate Before or After 4 Days of Ketogenic Diet
Time Frame: At baseline (approximatively 1 month before the onset of the diet) and right after a 4 days ketogenic diet
Measure: Mean (Standard Error); unit: µmol/100g/min
Groups:
- Ketogenic Diet: TEP study with a 4 days ketogenic diet
  Ketogenic diet: 4 days 4:1 (lipids:protein/carbohydrates) ketogenic diet
  Intervention 1: Pre-KD = Participants did a TEP before starting 4 days of ketogenic diet
  Intervention 2: Post-KD = Participants did a TEP after 4 days of ketogenic diet
Arm/Group | Ketogenic Diet
Number analyzed (Participants) | 10
µmol/100g/min
  Pre-KD | 0.672 (0.18)
  Post-KD | 4.83 (0.75)

2. Primary Outcome: Mean in Cerebral Metabolic Rate of Glucose Before or After 4 Days of Ketogenic Diet
Time Frame: At baseline (approximatively 1 month before the onset of the diet) and right after a 4 days ketogenic diet
Measure: Mean (Standard Error); unit: µmol/100g/min
Groups:
- Ketogenic Diet: TEP study with a 4 days ketogenic diet
  Ketogenic diet: 4 days 4:1 (lipids:protein/carbohydrates) ketogenic diet
Arm/Group | Ketogenic Diet
Number analyzed (Participants) | 10
µmol/100g/min
  Pre-KD | 31.58 (3.02)
  Post-KD | 24.46 (5.47)

ADVERSE EVENTS:
Groups:
- Ketogenic Diet: TEP study with a 4 days ketogenic diet
  Ketogenic diet: 4 days 4:1 (lipids:protein/carbohydrates) ketogenic diet
  Intervention 1: Pre-KD = Participants did a TEP before starting a 4 days ketogenic diet Intervention 2: Post-KD = Participants did a TEP after 4 days of ketogenic diet
Arm/Group | Ketogenic Diet
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes